CLINICAL TRIAL: NCT05483387
Title: Prospective Post-market Clinical Follow-up Study of the HBS 2 Resorb Mg in Patients With Intra- and Extraarticular Fractures, Pseudarthroses and Arthrodesis of Small Bones and Bone Fragments.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KLS Martin (Industry)
Collaborators: Clinical Study Centers, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMCF-00007_PLAN_002
Record Dates: First submitted 2022-07-28; First posted 2022-08-02 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Intraarticular Fracture; Extraarticular Fracture; Pseudarthrosis; Arthrosis
Keywords: small Bone; resorbable Implant; Magnesium
MeSH Terms: conditions — Intra-Articular Fractures; Pseudarthrosis; Osteoarthritis | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBS 2 Resorb Mg (Experimental): Study arm treated with the HBS 2 Resorb Mg.
  Interventions: Device: Treatment with HBS 2 Resorb Mg

INTERVENTIONS:
Device: Treatment with HBS 2 Resorb Mg — Treatment of fractures, arthrodesis or pseudarthroses of small bones and bone fragments

SUMMARY:
This study is a multi-centre, prospective, clinical observational study to evaluate the CE-marked HBS 2 Resorb Mg screws under routine conditions. The device will be used according to its intended use. The data collected for this study does only include measurements which are standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years and older
* Patient is undergoing surgery with HBS 2 Resorb Mg
* Written informed consent obtained for the treatment
* Treatment of intra-articular and extra articular fractures and pseudarthroses of small bones and bone fragments as well as arthrodeses in the treatment of:
* Scaphoid fractures and scaphoid pseudarthroses
* Proximal radius head fractures
* Fractures of the radial styloid process
* Fractures of the ulnar styloid process
* Metacarpal fractures
* Metatarsal fractures

Exclusion Criteria:

* Any not medically managed severe systemic disease
* Recent history of substance abuse (i.e. recreational drugs, alcohol) that would preclude reliable assessment
* Pregnancy or women planning to conceive within the study period
* Persons who are legally detained in an official institution
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study
* Skeletally immature
* Intraoperative decision to use implants other than the device under investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Bony Fusion (Change) | 6 weeks, 12 weeks, 6 month and 12 month after surgery
  The primary endpoint of the study is the fusion rate of the bone. After the onset of bony fusion, the implant no longer fulfils any function, and it should be resorbed.

SECONDARY OUTCOMES:
Secondary displacement and breakage of the implant (YES/NO) | 6 weeks, 12 weeks, 6 month and 12 month after surgery
  Any secondary radiographic displacement or breakage of the implant or any clinically significant loss of reduction is noted.
Deep infection(YES/NO) | 6 weeks, 12 weeks, 6 month and 12 month after surgery
  The presence of deep infections is assessed binary.
Clinical outcome | 6 weeks, 12 weeks, 6 month and 12 month after surgery
  Patient pain (VAS) and outcome measures (Patient Related Outcome Measure) will be noted in order to assess patient satisfaction.
Surgical revisions(YES/NO) | 6 weeks, 12 weeks, 6 month and 12 month after surgery
  As typically one single surgery should be sufficient to treat the patient, all secondary surgical interventions are revisions due to a complication. This includes also re-operation due to screw removal.
Early corrosion phenomenon(YES/NO) | 6 weeks, 12 weeks, 6 month and 12 month after surgery
  Symptomatic gas accumulation or formation of gas pockets due to degradation of the material.
Radiolucency(YES/NO) | 6 weeks, 12 weeks, 6 month and 12 month after surgery
  Any radiolucency on the postoperative X-rays are noted. Radiolucency will be assessed by the operating surgeon.

CONTACTS AND LOCATIONS:
Locations (1):
- Centrum für Muskuloskeletale Chirurgie (CMSC), Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided